CLINICAL TRIAL: NCT04916145
Title: A Single-center, Randomized, Open Label, No-treatment Controlled, Digital Device Study to Evaluate the Efficacy, Safety and Feasibility of SAT-008 in Healthy Adults
Brief Title: An Investigator-initiated, Explorative Trial Evaluating the Effect of SAT-008 in Healthy Adults
Acronym: SAT-008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Korea University Guro Hospital (Other); S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Yoon-Seok Chang, MD, PhD, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-2009-637-306
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Allergy and Immunology
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two study arms. One group (treatment) will receive an experimental digital device for 13 weeks while the other group (control) will maintain daily activity as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No any treatment (No Intervention): Participants randomly assigned to this group will maintain a routine life without any treatments (no use of SAT-008).
- Use of SAT-008 (Experimental): Participants randomly assigned to this group will be treated by SAT-008 during the study.
  Interventions: Device: SAT-008

INTERVENTIONS:
Device: SAT-008 — SAT-008 is a digital device containing several types of activities related to the immune function of adults.
  Arms: Use of SAT-008

SUMMARY:
The purpose of this exploratory study is to evaluate the efficacy, safety, and feasibility of a novel digital device called SAT-008 in healthy adults.

DETAILED DESCRIPTION:
This clinical study was designed as a single institution, open, controlled, and investigator-led clinical trial to evaluate the efficacy, safety, and feasibility of a novel digital device called SAT-008 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 50 years
* Received influenza vaccination the previous year
* Scheduled to receive the influenza vaccine
* Voluntarily agrees with a consent form

Exclusion Criteria:

* Current infectious disease
* History of autoimmune diseases
* Current immunological compromised diseases.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Changes in functions of immunocytes | Baseline, Week 1, Week 5, Week 13
  To measure changes in functions of natural killer cells, T cells, and B cells at 1, 5, and 13 weeks compared to baseline.
Number of expected and unexpected adverse events | Baseline
  To evaluate the safety of SAT-008
Number of expected and unexpected adverse events | Week 1 (a week following baseline)
  To evaluate the safety of SAT-008
Number of expected and unexpected adverse events | Week 5 (five weeks following baseline)
  To evaluate the safety of SAT-008
Number of expected and unexpected adverse events | Week 13 (thirteen weeks following baseline)
  To evaluate the safety of SAT-008
Rate of adherence to SAT-008 | Week 1 (a week following baseline)
  To assess a degree to which participants follow SAT-008
Rate of adherence to SAT-008 | Week 5 (five weeks following baseline)
  To assess a degree to which participants follow SAT-008
Rate of adherence to SAT-008 | Week 13 (thirteen weeks following baseline)
  To assess a degree to which participants follow SAT-008

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Seok Chang, MD, PhD, Principal Investigator — addchang@snu.ac.kr
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi JP, Ayoub G, Ham J, Huh Y, Choi SE, Hwang YK, Noh JY, Kim SH, Song JY, Kim ES, Chang YS. Exercise With a Novel Digital Device Increased Serum Anti-influenza Antibody Titers After Influenza Vaccination. Immune Netw. 2023 Feb 27;23(2):e18. doi: 10.4110/in.2023.23.e18. eCollection 2023 Apr. PMID 37179746